CLINICAL TRIAL: NCT01964820
Title: Online Positive Emotion Skills Intervention for Symptoms of Depression - Pilot Feasibility Trial
Brief Title: Online Positive Emotion Skills Intervention for Symptoms of Depression
Acronym: MARIGOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCSF CHR 13-12256
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Depression; Psychological Stress; Affect
MeSH Terms: conditions — Depression; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive affect skills intervention (Experimental): Participants receive a 5-week intervention providing training in 8 skills for generating positive affect.
  Interventions: Behavioral: Positive Affect Skills Training
- Emotion reporting (No Intervention): Participants report emotions on the same regular basis as intervention participants, but receive no intervention.

INTERVENTIONS:
Behavioral: Positive Affect Skills Training — Our intervention teaches 8 skills that research suggests lead to increased positive emotions, beginning with basic skills (recognizing and savoring positive events), and progressing to more complex ones such as goal- setting and acts of kindness. Established skills such as reappraising negative thoughts are also taught, in the context of cultivating positive emotions and coping with stress.
  The skills are taught over 5 weeks, with one or more new skills introduced each week. A week consists of 1-2 days of didactic material and 5-6 days of real-life skills practice and reporting.
  For a full description, see "A positive affect intervention for people experiencing health-related stress: development and non-randomized pilot test" (Moskowitz et al., 2012).
  Other Names: DAHLIA; MARIGOLD
  Arms: Positive affect skills intervention

SUMMARY:
Major depressive disorder affects over 120 million people worldwide. Only 50% of Americans with depression receive adequate treatment, and one-third of those receiving treatment do not benefit. In this pilot project investigators will bring together two approaches that have the promise to reach large numbers of depression sufferers: a skills-based intervention for increasing positive affect and experiences in depressed individuals, delivered in an inexpensive self-paced mobile format. The study will make use of smartphone technology to improve conventional outcome measurement via in-the-moment emotion sampling and mobile assessment of heart rate variability, a predictor of cardiac health that may mediate some of the health effects of depression. The aims are: 1) Retool the existing web-based positive emotion intervention for use on smartphones, with innovative exercises that help participants bring the skills they are learning into real- life situations; 2) Measure heart rate variability and emotions using existing smartphone software; and 3) Perform a randomized pilot trial of the mobile intervention on individuals with clinical depression recruited online.

ELIGIBILITY:
Inclusion Criteria:

* Daily internet access
* Cell phone ownership
* Score of 10 or greater on the PHQ-8 depression scale

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Retention / feasibility | 3 months after completion of intervention (5 months post-enrollment, may be slightly more or less for intervention participants depending on time taken to complete the course)
  Determine percentage of participants providing data at each stage of the study (intervention phase, post-intervention, 1 month followup, 3 month followup)
Depression symptoms (PHQ-9 questionnaire) | 60 days after enrollment (administered immediately post-intervention, may be slightly more or less than 60 days for intervention participants depending on time taken to complete the course)
Depression symptoms (CES-D questionnaire) | 60 days after enrollment (administered immediately post-intervention, may be slightly more or less than 60 days for intervention participants depending on time taken to complete the course)

SECONDARY OUTCOMES:
Perceived Stress (PSS questionnaire) | 60 days after enrollment (administered immediately post-intervention, may be slightly more or less than 60 days for intervention participants depending on time taken to complete the course)
Positive and Negative affect (DES questionnaire) | 60 days after enrollment (administered immediately post-intervention, may be slightly more or less than 60 days for intervention participants depending on time taken to complete the course)
Depression symptoms at follow-up (CESD questionnaire) | 3 months after completion of intervention (5 months post-enrollment, may be slightly more or less for intervention participants depending on time taken to complete the course)
Depression symptoms at follow-up (PHQ-9 questionnaire) | 3 months after completion of intervention (5 months post-enrollment, may be slightly more or less for intervention participants depending on time taken to complete the course)

CONTACTS AND LOCATIONS:
Overall Officials: Judith T Moskowitz, PhD, Principal Investigator — University of California, San Francisco; Michael A Cohn, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco - Osher Center for Integrative Medicine, San Francisco, California, United States

REFERENCES:
- [Background] Moskowitz JT, Hult JR, Duncan LG, Cohn MA, Maurer S, Bussolari C, Acree M. A positive affect intervention for people experiencing health-related stress: development and non-randomized pilot test. J Health Psychol. 2012 Jul;17(5):676-92. doi: 10.1177/1359105311425275. Epub 2011 Oct 21. PMID 22021272
- [Derived] Cheung EO, Addington EL, Bassett SM, Schuette SA, Shiu EW, Cohn MA, Leykin Y, Saslow LR, Moskowitz JT. A Self-Paced, Web-Based, Positive Emotion Skills Intervention for Reducing Symptoms of Depression: Protocol for Development and Pilot Testing of MARIGOLD. JMIR Res Protoc. 2018 Jun 5;7(6):e10494. doi: 10.2196/10494. PMID 29871853